CLINICAL TRIAL: NCT02889328
Title: Phase II Study of Continuous Dosing of Regorafenib in Patients With Gastrointestinal Stromal Tumors (GISTs) After Failure of Imatinib and Sunitinib: GIST Regorafenib Continuous Dosing
Brief Title: Phase II Study of Regorafenib Continuous Dosing of Regorafenib in Patients With GISTs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC1602
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Gastrointestinal Stromal Tumors (GISTs)
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- regorafenib (Experimental): regorafenib 100 mg po od daily, every 4 weeks (28 day)
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — Regorafenib 100mg continuous dosing arm

SUMMARY:
Randomized, placebo-controlled, phase III study of regorafenib 160 mg once daily on intermittent dosing schedule of 3 weeks on treatment followed by 1 weeks off demonstrated the significant benefit of regorafenib in terms of PFS in patients with GISTs who had failed to both imatinib and sunitinib. However, there are concerns that tumors and tumor-related symptoms may be progressed during off treatment period. Investigators hypothesize that continuous dosing schedule of regorafenib might be feasible and effective to prevent disease flare on off-treatment period. Based on the results of previous dose escalation study for continuous regorafenib dosing, we investigate the 100 mg daily dose of regorafenib in patients with TKI-refractory GISTs.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 years or older, at the time of acquisition of informed consent
* Histologically confirmed metastatic and/or advanced (unresectable or recurrent) GIST with CD117(+), DOG-1(+), or mutation in KIT or PDGFRα gene
* Disease progression or intolerance to imatinib as well as disease progression on sunitinib Disease progression is defined as (1) size increase > 20% by RECIST version 1.1, (2) appearance of a definite new lesion (excluding small cystic new lesions in the liver within 6 months of starting TKIs), (3) new solid nodule within a cystic mass, or (4) increase of the size (> 20%) of previously existing solid nodule within a cystic mass. Intolerance to previous TKIs is defined as (1) drug compliance < 75% due to grade 2 or more non-hematologic toxicities despite dose reduction to one dose level below (300 mg per day for imatinib; 37.5 mg per day on a 4 weeks on and 2 weeks off schedule or 25 mg per day continuous dosing for sunitinib), (2) Febrile neutropenia, grade 4 neutropenia for more than 6 days, grade 4 thrombocytopenia, grade 3 thrombocytopenia with clinically significant bleeding, grade 3-4 or continuous intolerable grade 2 non-hematologic toxicities despite dose reduction to one dose level below as described above.
* ECOG performance status of 0~1
* Resolution of all toxic effects of prior treatments to grade 0 or 1 by NCI-CTCAE version 4.03
* At least one measurable lesion as defined by RECIST version 1.1.
* Adequate bone marrow, hepatic, renal, and other organ functions
* Neutrophil > 1,500/mm3
* Platelet > 100,000/mm3
* Hemoglobin > 9.0 g/dL
* Total bilirubin < 1.5 x upper limit of normal (ULN)
* Lipase ≤ 1.5 x the ULN
* AST/ALT < 3.0 x ULN (or < 5 x ULM in case of liver metastases)
* Alkaline phosphatase (ALP) limit ≤ 2.5 x ULN (≤5 x ULN for patients with liver involvement of their cancer and /or have bone metastases).
* Estimated creatinine clearance (CLcr) ≥ 30 mL/min as calculated using the Cockcroft-Gault equation.
* International normalized ratio (INR) ≤ 1.5 x ULN and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless receiving treatment with therapeutic anticoagulation. Patients being treated with anticoagulant, e.g. heparin, will be allowed to participate provided no prior evidence of an underlying abnormality in these parameters exists. Close monitoring of at least weekly evaluations will be performed until INR and PTT are stable based on a pre-dose measurement as defined by the local standard of care.
* Electrolytes should be within normal limits.
* Urine dipstick reading: Negative for proteinuria or, if documentation of +1 results for protein on dipstick reading, then total urinary protein ≤ 500 mg and measured creatinine clearance ≥ 30 mL/min/1.73m2 from a 24-hour urine collection
* Life expectancy > 12 weeks
* Women with reproductive potential must have a negative serum or urine pregnancy test; and men and women of reproductive potential must practice an effective method of avoiding pregnancy while receiving study drug.
* Provision of a signed written informed consent
* Women of childbearing potential and men must agree to use adequate contraception before entering the program until at least 8 weeks after the last study drug administration. The investigator or a designated associate is requested to advise the subject on how to achieve an adequate birth control. Adequate contraception is defined in the study as any medically recommended method (or combination of methods) as per standard of care
* Women of childbearing potential must have a blood or urine pregnancy test performed a maximum of 7 days before start of study treatment, and a negative result must be documented before start of study treatment

Exclusion Criteria:

* Prior use of any VEGFR inhibitor other than sunitinib (e.g., sorafenib)
* Subjects who have received:

-any other approved tyrosine kinase inhibitor within 1 week or a minimum 5 drug half- lives, whichever is longer (i.e., within 7 days for imatinib or within 10 days for sunitinib)

* any other investigational new drugs within 4 weeks or 5 drug half-lives (if drug half-life in subjects is known), whichever is shorter.

  * Women of child-bearing potential who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control.
  * Clinically significant cardiac disease (New York Heart Association, Class III or IV) or impaired cardiac function or clinically significant cardiac diseases, including any one of the following:
  * LVEF < 45% as determined by MUGA scan or echocardiogram
  * Complete left bundle branch block
  * Obligate use of a cardiac pacemaker
  * Congenital long QT syndrome
  * History or presence of ventricular tachyarrhythmia
  * Presence of unstable atrial fibrillation (ventricular response > 100 bpm). Patients with stable atrial fibrillation are eligible, provided they do not meet any of the other cardiac exclusion criteria
  * Clinically significant resting bradycardia (< 50 bpm)
  * Uncontrolled hypertension (systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 100 mmHg, with or without anti-hypertensive medication).
  * QTc > 480 msec on screening ECG
  * Right bundle branch block + left anterior hemiblock (bifasicular block)
  * Angina pectoris ≤ 3 months prior to starting study drug
  * Acute Myocardial Infarction ≤ 3 months prior to starting study drug
  * Other clinically significant heart disease (e.g., CHF, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
  * Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
  * Diabetes mellitus (insulin dependent or independent disease, requiring chronic medication) with signs of clinically significant peripheral vascular disease.
  * Previous pericarditis; clinically significant pleural effusion in the previous 12 months or current ascites requiring two or more interventions/month.
  * Known pre-existing clinically significant disorder of the hypothalamic-pituitary axis, adrenal or thyroid glands.
  * Prior acute or chronic pancreatitis of any etiology.
  * Acute and chronic liver disease and all chronic liver impairment.
  * Malabsorption syndrome or uncontrolled gastrointestinal toxicities (nausea, diarrhea, vomiting) with toxicity greater than NCI CTCAE grade 2.
  * Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for this study.
  * Treatment with any of the medications that have a potential risk of prolonging the QT interval or inducing Torsades de Points and the treatment cannot be discontinued or switched to a different medication prior to starting study drug.
  * Use of ketoconazole, erythromycin, carbamazepine, phenobarbital, rifampin, phenytoin and quinidine 2 weeks prior baseline.
  * Major surgery ≤ 28 days prior to starting study drug or who have not recovered from side effects of such therapy.
  * Known diagnosis of HIV infection (HIV testing is not mandatory).
  * History of another primary malignancy that is currently clinically significant or currently requires active intervention.
  * Patients with brain metastases as assessed by radiologic imaging (e.g. CT, MRI)
  * Alcohol or substance abuse disorder.
  * Non-healing wound, non-healing ulcer, or non-healing bone fracture
  * Patients with evidence or history of any bleeding diathesis, irrespective of severity
  * Any hemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to the start of study medication.
  * Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 month before the start of study medication (except for adequately treated catheter-related venous thrombosis occurring more than one month before the start of study medication)
  * Active hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy.
  * Ongoing infection > Grade 2 NCI CTCAE

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-09; Primary Completion 2017-08-09 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Disease control rate | at least 12 weeks
  Disease control rate (CR + PR + SD) lasting for at least 12 weeks according to the RECIST v1.1

SECONDARY OUTCOMES:
Progression-free survival | up to 2 years
Overall survival | up to 2 years
Toxicity profile by the NCI-CTCAE v4.03 | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim JJ, Ryu MH, Yoo C, Beck MY, Ma JE, Kang YK. Phase II Trial of Continuous Regorafenib Dosing in Patients with Gastrointestinal Stromal Tumors After Failure of Imatinib and Sunitinib. Oncologist. 2019 Nov;24(11):e1212-e1218. doi: 10.1634/theoncologist.2019-0033. Epub 2019 Apr 29. PMID 31036770